# 16.1.9 Documentation of Statistical Methods

- 16.1.9.1 Statistical Analysis Plan
- **16.1.9.2 MiniSim Drive Summary Measures**

# 16.1.9.1 Statistical Analysis Plan

The Statistical Analysis Plan dated 13 October 2017 is attached.

### STATISTICAL ANALYSIS PLAN

**PROTOCOL: 115** 

# Driving Simulation Cross-Over Study of Sedative Effects of Tolperisone Compared to Cyclobenzaprine and Placebo

**SPONSOR:** Neurana Pharmaceuticals, Inc.

3525 Del Mar Heights Rd, #609

San Diego, CA 92130

**PRODUCT:** Tolperisone hydrochloride, NR100

**AUTHOR:** Jeffrey S Finman, PhD

Jupiter Point Pharma Consulting, LLC

796 Shennecossett Road

Groton, CT 06340

Julie M Jones, PhD

Breckenridge Statistics, Inc. 226 S Main St. Unit 20

PO Box 1849

Breckenridge, CO 80424

**DATE:** October 13, 2017

**STATUS:** Final Version 1.0

# Statistical Analysis Plan

Protocol: 115

Final Version: 1.0 Date: 13-Oct-2017

| CRO | REPRESENTATIV | E |
|---|---|---|
| | VIEWED AND APP | PROVED BY: |
| SIGNATURE: | 145/ | DATE: 17 OCT 201 |
| NAME: Gary Kay PhD. | _ · / | |
| DEPARTMENT/TITLE: President Cogniti | ve Research Corpora | ndon |
| STATISTIC | AL CRO REPRESEN | VIATIVE |
| | VIEWED AND APP | |
| SIGNATURE TILLE | | DATE: 170072017 |
| NAME: Julie Jones PhD. | | 10012011 |
| DEPARTMENT/TITLE: President, Brecke | and described to | |
| Det in the interest of the int | mage Statistics inc. | |
| STATISTICA | AL CRO REPRESEN | TATIVE |
| DOCUMENT RE | VIEWED AND APP | ROVED BY: |
| SIGNATURE: | - rain | DATE: 12-0ct-2017 |
| NAME: Jeffrey Finman PhD. | | 17-04-2011 |
| DEPARTMENT/TITLE: President, Jupiter | Point Consulting | |
| | 7-10-00-00-00 | · |
| SPONSO | OR REPRESENTAT | IVE |
| DOCUMENT RE | VIEWED AND APP | ROVED BY: |
| SIGNATURE: SCALOR | | DATE:/0/13/17 |
| NAME: Judy Caron PhD. | | |
| DEPARTMENT/TITLE: Chief Operating O. | fficer Neuman Phare | macartinela |

### **TABLE OF CONTENTS**

| 1 | LIST OF ABBREVIATIONS | 5 |
|---|---|---|
| 2 | INTRODUCTION | 6 |
| 3 | | |
| J | | |
| | 3.1 PRIMARY OBJECTIVE | |
| 4 | STUDY DESIGN | |
| 4 | | |
| | <ul><li>4.1 DURATION OF STUDY</li></ul> | 6 |
| | 4.3 DESIGN AND TREATMENTS | 6 |
| _ | ABLE 1 SCHEMATIC OF DESIGN | |
| ı | | |
| | 4.4 TREATMENTS | |
| | 4.4.1 Tolperisone Dose Level | |
| | 4.5 RANDOMIZATION | |
| | 4.5.1 SCHEDULE OF EVENTS AND ASSESSMENTS | 9 |
| т | ABLE 2 SCHEDULE OF ACTIVITIES | 10 |
| 5 | OUTCOME VARIABLE DEFINITIONS | 12 |
| | 5.1 SCREENING AND BASELINE ASSESSMENT | |
| | 5.2 PHARMACODYNAMIC ASSESSMENTS | |
| | 5.2.1 CVDA DRIVING SCENARIO ON THE CRCDS-MiniSim | |
| | 5.2.2 KAROLINSKA SLEEPINESS SCALE (KSS) | 12 |
| | 5.2.3 SELF PERCEIVED SAFETY TO DRIVE QUESTION | |
| | 5.2.4 COGSCREEN SYMBOL DIGIT CODING (SDC) | 13 |
| | 5.2.5 VISUAL ANALOG SCALE (VAS) TO ASSESS MOTIVATION AND SELF-APPRAISAL 5.3 PHARMACODYNAMIC ENDPOINTS | 13 |
| | 5.3.1 PRIMARY ENDPOINT | |
| | 5.3.2 SECONDARY ENDPOINTS | |
| | 5.4 SAFETY ASSESSMENTS | |
| | 5.4.1 SECONDARY SAFETY ENDPOINTS | |
| | 5.4.2 ADVERSE EVENTS | |
| | 5.4.3 CLINICAL LABORATORY EVALUATIONS | 15 |
| | 5.4.4 PHYSICAL EXAMINATION | |
| | 5.4.5 VITAL SIGNS | 16 |
| | 5.4.6 12-LEAD ELECTROCARDIOGRAM | |
| | 5.5 CONCOMITANT MEDICATIONS | |
| | 5.6 SCREENING ASSESSMENTS | |
| | 5.6.1 EPWORTH SLEEPINESS SCALE | 17 |
| 6 | STATISTICAL ANALYSES | 17 |
| | 6.1 STATISTICAL METHODOLOGY | 17 |
| | 6.1.1 DETERMINATION OF SAMPLE SIZE | |
| | 6.1.2 ANALYSIS POPULATIONS | |
| | 6.1.3 STATISTICAL ANALYSES – GENERAL CONSIDERATIONS | |
| | 6.1.4 MULTIPLE COMPARISONS | 18 |
| | 6.1.5 PROCEDURES FOR HANDLING MISSING DATA | 19 |

| 6.2 SCREENING AND BASELINE CHARACTERISTICS | 18 |
|--------------------------------------------|------------|
| 6.3 SUBJECT DISPOSITION | 19 |
| 6.4 STUDY MEDICATION ADMINISTRATION | 20 |
| 6.5 PHARMACODYNAMIC ANALYSES | |
| 6.5.1 PRIMARY ANALYSIS | 20 |
| 6.5.2 SECONDARY ANALYSES | 21 |
| 6.6 SAFETY ANALYSES | |
| 6.6.1 ADVERSE EVENTS (AE) | |
| 6.6.2 CLINICAL LABORATORY EVALUATIONS | 23 |
| 6.6.3 PHYSICAL EXAMINATION | |
| 6.6.4 VITAL SIGNS | 23 |
| 6.6.5 12-LEAD ELECTROCARDIOGRAM | |
| 6.7 CONCOMITANT MEDICATIONS | 24 |
| 6.8 CONCENTRATION DATA | 24 |
| 6.9 ADDITIONAL COLLECTED DATA | 24 |
| 7 REFERENCES | <b>2</b> 4 |
| 8 TABLES, LISTINGS, AND FIGURES | 25 |
| 8.1 TABLES | 25 |
| 8.2 LISTINGS | |
| 8.3 FIGURES | |

# 1 LIST OF ABBREVIATIONS

| AE(s) | Adverse event(s) |
|---------------|----------------------------------------------------------|
| BAC | Blood Alcohol Content |
| BMI | Body mass index |
| CRCDS-MiniSim | Cognitive Research Corporation Driving Simulator-MiniSim |
| CRF | Case report form |
| CVDA | Country Vigilance-Divided Attention |
| DA | Divided attention |
| ECG | Electrocardiogram |
| EOS | End of study |
| ESS | Epworth Sleepiness Scale |
| HIV | Human immunodeficiency virus |
| ITT | Intent-to-Treat |
| KSS | Karolinska Sleepiness Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mm | Millimeter |
| N | Number |
| NI | Non-inferiority |
| PK | Pharmacokinetic |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SDC | Symbol Digit Coding |
| SDLP | Standard deviation of lateral position |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TID | Three times a day |
| VAS | Visual analog scale |

#### 2 INTRODUCTION

This statistical analysis plan (SAP) describes the planned statistical analyses for the study entitled "Driving Simulation Cross-Over Study of Sedative Effects of Tolperisone Compared to Cyclobenzaprine and Placebo" finalized 28 April 2017.

#### 3 STUDY OBJECTIVE

#### 3.1 PRIMARY OBJECTIVE

The primary objective of this study is:

to assess the sedative effect of 150 mg TID tolperisone and 10 mg TID cyclobenzaprine compared to placebo on simulated driving performance and cognitive functioning in healthy adult volunteers. In this crossover study, treatment effects will be assessed following the second initial dose, the morning following nighttime dosing (to assess residual next day effects), and at steady state (i.e., following AM dosing on Day 3).

#### 3.2 SECONDARY OBJECTIVE

The secondary objective of this study is:

 to assess the safety of 150 mg TID tolperisone dosing for 3 days in healthy volunteers.

#### 4 STUDY DESIGN

#### 4.1 DURATION OF STUDY

The total duration of study participation will be approximately 4 weeks (range 4-8 weeks), including Screening and Follow-up. Subject participation will be approximately 3 weeks as outpatients with 3 days each week as overnight clinic participants.

#### 4.2 NUMBER OF SUBJECTS (STUDY POPULATION)

A sufficient number of subjects will be enrolled to ensure a total of 30 normal, healthy, male and female subjects between the ages of 21 and 55 years (at the time of informed consent) will complete all dosing periods, including the driving assessment.

#### 4.3 DESIGN AND TREATMENTS

This will be a randomized, placebo-controlled, multiple-dose 3-way cross-over study of the safety and cognitive effects of multiple doses of tolperisone administered TID in 30 male and female healthy volunteers. Treatment groups include 450 mg tolperisone (i.e., 150 mg administered three times daily), 30 mg cyclobenzaprine (i.e., 10 mg administered three times daily), and placebo.

Subjects will be dosed on the morning of Day 1. Approximately one hour after the second dose on Day 1, subjects will be administered the cognitive test, followed by the driving simulator examination.

On the morning of Day 2, prior to dosing, subjects will be readministered the cognitive test and driving examination to assess residual next day effects.

Subjects will repeat cognitive testing and the driving examination on the morning of Day 3, after administration of the AM study medication, to evaluate the cumulative effects of 3 days of dosing.

Subjects will be discharged on Day 3 with instructions to return to the clinic on Day 7 and Day 14 to repeat the above procedures with the second and third treatments.

A follow-up phone call will be conducted 1 week (±3 days) following discharge from the clinic on Day 17 to assess for continued safety.

A schematic of the study design is presented in <u>Table 1</u>.

Table 1 Schematic of Design



#### 4.4 TREATMENTS

#### 4.4.1 Tolperisone Dose Level

For the tolperisone treatment arm, tolperisone will be administered three times per day, with 1 tablet administered at 8:00 AM (AM dose), 2:00 PM (PM dose), and 10:00 PM (HS dose) daily for 2 days and 1 tablet at 8:00 AM on Day 3. Depending upon randomization sequence tolperisone dosing will take place at Visit 1, 2, or 3. Each dose will be a 150 mg tablet of tolperisone, for a total daily dose of 450 mg on Days 1 and 2, and a total dose of 150 mg on Day 3.

#### 4.4.2 Positive Control Dose Level

Cyclobenzaprine will serve as the positive control to demonstrate assay sensitivity. For the cyclobenzaprine treatment arm, cyclobenzaprine will be administered three times per day, with 1 tablet administered at 8:00 AM (AM dose), 2:00 PM (PM dose), and 10:00 PM (HS dose) daily for 2 days and 1 tablet at 8:00 AM on Day 3. Depending upon randomization sequence, cyclobenzaprine dosing will take place at Visit 1, 2, or 3. Each dose will be a 10

mg tablet of cyclobenzaprine, for a total daily dose of 30 mg on Days 1 and 2, and a total dose of 10 mg on Day 3.

#### 4.5 RANDOMIZATION

Prior to dosing, subjects will be randomly assigned to one of 6 treatment sequences (one for each permutation of treatment groups) and dosed with study medication (tolperisone, cyclobenzaprine or placebo) based upon a randomization scheme provided by Cognitive Research Corporation. Only the qualified person(nel) assigned to prepare and administer the study treatment will have access to the randomization schedule and dispensing records during the study period.

#### 4.5.1 SCHEDULE OF EVENTS AND ASSESSMENTS

The schedule of study events and assessments are presented in <u>Table 2</u>.

**Table 2 Schedule of Activities** 

| | Screenin Period 1 | | | | | Period 2 | | | | Period 3 | | | | Follow-up<br>Phone<br>Call |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Day -28<br>to -2<br>(V1) | Day -1<br>(V2) | Day 1<br>(V3) | Day 2<br>(V4) | Day 3<br>(V5) | Day 7<br>(V6) | Day 8<br>(V7) | Day 9<br>(V8) | Day 10<br>(V9) | Day 14<br>(V10) | Day 15<br>(V11) | Day 16<br>(V12) | Day 17<br>(V13) | Day 24<br>(±3 days)<br>(V14) |
| Informed Consent | х | | | | | | | | | | | | | |
| Inclusion/Exclusion Review | Х | х | | | | Х | | | | Х | | | | |
| Medical/Social History | Х | | | | | | | | | | | | | |
| Physical Examination | Х | | | | | | | | | | | | Х | |
| Epworth Sleepiness Scale | Х | | | | | | | | | | | | | |
| Simulator Sickness<br>Questionnaire | Х | | | | | | | | | | | | | |
| Driving Simulation & Cognitive Testing practice | Х | Х | | | | х | | | | Х | | | | |
| Driving Simulation & Cognitive Testing | | | х | х | x | | х | Х | Х | | Х | Х | Х | |
| KSS | | | Х | Х | Х | | Х | Х | Х | | Х | Х | Х | |
| Self-Perceived<br>Questionnaire | | | х | х | Х | | х | Х | х | | х | Х | Х | |
| VAS | | | Х | Х | Х | | Х | Х | Х | | Х | Х | Х | |
| Vital Sign Measurements <sup>a</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Standard 12-Lead ECG | Х | | | | | | | | | | | | Х | |

| | Screenin<br>g | Period 1 | | | Period 2 | | | Period 3 | | | | Follow-up<br>Phone<br>Call | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Day -28<br>to -2<br>(V1) | Day -1<br>(V2) | Day 1<br>(V3) | Day 2<br>(V4) | Day 3<br>(V5) | Day 7<br>(V6) | Day 8<br>(V7) | Day 9<br>(V8) | Day 10<br>(V9) | Day 14<br>(V10) | Day 15<br>(V11) | Day 16<br>(V12) | Day 17<br>(V13) | Day 24<br>(±3 days)<br>(V14) |
| Laboratory Evaluations <sup>b</sup> | Х | | | | | | | | | | | | Х | |
| Serum/Urine Pregnancy<br>Test <sup>c</sup> | х | Х | | | | х | | | | Х | | | | |
| Urine Drug Screening /<br>Breathalyzer | х | Х | | | | х | | | | Х | | | | |
| Pharmacokinetic Sampling <sup>d</sup> | | | Х | Х | Х | | Х | Х | Х | | Х | Х | Х | |
| Adverse Events | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| Concomitant Medications | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| Study Drug Administration | | | Х | Х | Х | | Х | Х | Х | | Х | Х | Х | |
| Discharge from Clinic | | | | | Х | | | | Х | | | | Х | |

a Vital signs include supine and standing blood pressure and heart rate; respiration rate; and body temperature. Weight and height collected at Visit 1 only.

b Laboratory Evaluations include hematology, serum chemistry, and urinalysis.

A serum pregnancy test will be performed at Screening and a urine pregnancy test will be performed upon each admission to the unit. Blood samples for the determination of plasma tolperisone concentrations will be drawn prior to each AM dosing on Days 1-3 and post-driving test (15-30 minutes after the drive) on Days 1 and 3

#### 5 OUTCOME VARIABLE DEFINITIONS

#### 5.1 SCREENING AND BASELINE ASSESSMENT

#### Screening:

Demographic characteristics of age, sex, race, ethnicity, height, weight, and body mass index (BMI), informed consent, substance use (social history), inclusion criteria, exclusion criteria, medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), laboratory results, urine drug screen, alcohol screen, pregnancy test, Epworth Sleepiness Scale (ESS), CogScreen Training and practice, driving simulator training and practice, simulator sickness questionnaire, prior medications, and concomitant medications will be collected at Screening.

#### **Baseline Assessment:**

Eligibility, vital signs, urine drug screen, alcohol screen, pregnancy test, pharmacokinetic sampling, CogScreen practice, driving simulator practice, adverse events, and concomitant medications will be collected at Baseline.

#### 5.2 PHARMACODYNAMIC ASSESSMENTS

#### 5.2.1 CVDA DRIVING SCENARIO ON THE CRCDS-MiniSim

The present study employs the Cognitive Research Corporation Driving Simulator (CRCDS) Country Vigilance-Divided Attention (CVDA) driving scenario, a 62.1 mile (100 km), monotonous, two-lane highway driving task that includes a secondary visual vigilance task (Divided Attention DA). The monotonous Country Vigilance scenario has been demonstrated to be sensitive to detect the effects of fatigue or sleepiness on driving performance [CRCDS]. This scenario has been useful in measuring the effects of sleep deprivation, Obstructive Sleep Apnea, chronic primary insomnia, and is sensitive to central nervous system (CNS) depressants (e.g., alcohol and sedating antihistamines). Results obtained using this methodology are comparable to those obtained using over-the-road driving tests [Siemen, 2015].

Subjects will perform the driving simulator test at the times specified in <u>Table 2</u>. Data will be captured in electronic format. Details are provided in the Cognitive Research Corporation CRCDS Testing Operations Manual.

#### 5.2.2 KAROLINSKA SLEEPINESS SCALE (KSS)

The Karolinska Sleepiness Scale (KSS) (Akerstedt 1990) will be used to assess subjective level of sleepiness. This is a subject self-report measure of situational sleepiness and provides an assessment of alertness/sleepiness at a particular point in time. The KSS has been found to correlate with electroencephalogram and behavioral variables (Kaida 2006). It is a 9-point categorical Likert scale:

- (1) extremely alert
- (2)
- (3) alert
- (4)
- (5) neither sleepy nor alert
- (6)
- (7) sleepy but no difficulty remaining awake
- (8)
- (9) extremely sleepy-fighting sleep

#### 5.2.3 SELF PERCEIVED SAFETY TO DRIVE QUESTION

Prior to driving the subject will be asked a simple question as to whether they feel safe to drive ("Right now do you feel safe to drive?"). Subject will answer "yes" or "no".

#### 5.2.4 COGSCREEN SYMBOL DIGIT CODING (SDC)

The CogScreen Symbol Digit Coding (SDC) subtest will be used in this study to measure attention, visual scanning, working memory, and speed of information processing. SDC is a computer analogue of the conventional digit symbol substitution task found in the WAIS-R Digit Symbol subtest and the Symbol Digit Modalities Test (Wechsler 1981).

SDC will be administered by trained study site personnel. The subject will perform the test by interacting with a touchscreen monitor. Data will be captured in electronic format. Details are provided in the CogScreen® Examiner Manual, CogScreen LLC, 2016.

# 5.2.5 VISUAL ANALOG SCALE (VAS) TO ASSESS MOTIVATION AND SELF-APPRAISAL

After completing the driving simulation, subjects will assess their own performance and their level of motivation to perform at their best during the driving simulation.

Subjects will respond to 2 questions:

- 1. How well you think you drove for the last 60 minutes?
- 2. How motivated did you feel to drive at your best during the last 60 minutes of driving?

Subjects will record their response to each question by drawing a vertical line on a 100 mm horizontal, linear visual analog scale (VAS). For the self-assessment of driving performance, one end of the line is marked "Not Satisfactory" and the other end of the line is marked "Satisfactory". For the motivation item, one end of

the line is marked "Not Motivated" and the other end is marked "Motivated". Scores on the 100 mm linear scale will be measured to the nearest millimeter from the left. The subject's scores will be recorded in the case report form (CRF).

#### 5.3 PHARMACODYNAMIC ENDPOINTS

#### 5.3.1 PRIMARY ENDPOINT

The primary endpoint for this study is simulated driving performance as measured by standard deviation of lateral position (SDLP) using the CRCDS-MiniSim.

#### 5.3.2 SECONDARY ENDPOINTS

The secondary endpoints for this study are:

- SDLP
- KSS
- Self-reported readiness to drive ("Right now do you feel safe to drive?)
- VAS for motivation
- VAS for self-appraisal of driving performance
- SDC:
  - Number of correct responses
  - Accuracy
  - Standard deviation of reaction time
- Other Driving Performance Endpoints
  - o Lane exceedance; including number, maximum, and duration
  - Average speed, speed deviation, excessive speeding count, speeding ratio
  - Excessive Ay (cornering speed threshold exceeded)
  - Total collisions
  - DA measures: Correct Responses, Omission Errors, Commission Errors, Reaction Time, Standard Deviation of Reaction Time
- Plasma drug levels and driving performance

#### 5.4 SAFETY ASSESSMENTS

#### 5.4.1 SECONDARY SAFETY ENDPOINTS

The secondary safety endpoints for this study are:

- Adverse events (AEs)
- Laboratory safety tests (blood chemistry, hematology, urinalysis, serum and urine pregnancy tests for women of childbearing potential)
- Physical examinations
- Vital signs

- Orthostatic effects
- 12-lead electrocardiograms (ECGs)

#### 5.4.2 ADVERSE EVENTS

An AE is defined as any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. AEs occurring after the initiation of the treatment are referred to as treatment emergent adverse events (TEAEs). An AE can therefore be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. AEs will be captured from the time of obtaining informed consent until discharge from the study.

#### 5.4.3 CLINICAL LABORATORY EVALUATIONS

A certified laboratory will be used to perform all routine hematology, clinical chemistry, and urinalysis. Planned laboratory analyses include:

| Category | Test Name |
|------------|------------------------------------------------|
| Hematology | Hemoglobin |
| | Hematocrit |
| | Platelets |
| | Prothrombin Time <sup>c</sup> |
| | Red blood cells |
| | White blood cells with differential (absolute) |
| Chemistry | Alanine aminotransferase |
| | Aspartate aminotransferase |
| | Alkaline phosphatase |
| | Blood urea nitrogen |
| | Creatinine |
| | Gamma glutamyltransferase |
| | Glucose |
| | Potassium |
| | Sodium |
| | Total and direct bilirubin |
| | Thyroid stimulating hormone <sup>c</sup> |
| Urinalysis | Bilirubin |
| | Erythrocytes |
| | Glucose |
| | Ketones |
| | Leukocytes |
| | Nitrite |

Breckenridge Statistics, Inc.: Statistical Analysis Plan-Neurana 115 Draft Version 1.0

| Category | Test Name |
|----------|----------------------------------------------------|
| | pH |
| | Protein |
| | Specific gravity |
| | Urobilinogen |
| Other | Urine drug and alcohol breathalyzer <sup>a,b</sup> |
| | Serum/urine Pregnancy <sup>d</sup> |

- <sup>a</sup> Screening and end of study (EOS) (Day 17).
- b Includes testing for amphetamines, methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, ethanol and opiates – ethanol will be determined by breathalyzer.
- <sup>c</sup> Screening only.
- <sup>d</sup> Serum pregnancy at Screening and urine pregnancy test at check-in for each period (Days -1, 7, and 14) for females of childbearing potential.

Note: The complete panel of safety labs (other than where footnoted) will be completed at Screening and EOS (Day 17).

#### **5.4.4 PHYSICAL EXAMINATION**

A physical examination will be performed at Screening and End of Study (Day 17).

#### 5.4.5 VITAL SIGNS

Vital signs will include the measurement of supine and standing blood pressure and heart rate, respiration rate, and body temperature. Weight and height will be measured at Screening only.

Vital signs, including supine and standing blood pressure and heart rate, temperature and respiration rate will be collected at the following visits/time points:

- Screening,
- Day -1, 7, and 14 upon clinic check-in,
- Day 1, 2, 3, 8, 9, 10, 15, 16, and 17 prior to and 4 hours post AM dosing.

#### 5.4.6 12-LEAD ELECTROCARDIOGRAM

Twelve-lead ECG recording will be collected at Screening and End of Study (Day 17).

#### 5.5 CONCOMITANT MEDICATIONS

The use of any concomitant medication taken during the study, including any medication taken for the treatment of AEs, will be recorded in the case report form (CRF). Recording of a concomitant medication will include the medication name, indication, dose, route, frequency, date started and date stopped.

#### 5.6 SCREENING ASSESSMENTS

#### 5.6.1 EPWORTH SLEEPINESS SCALE

The Epworth Sleepiness Scale (ESS) will be used to exclude subjects who demonstrated excessive sleepiness prior to randomization.

The ESS is an 8-item self-administered questionnaire to measure general level of daytime sleepiness. The Scale is based on questions referring to situations that vary in their likelihood to induce a person to fall asleep. Subjects are asked to rate how likely they would be to doze off or fall asleep in each situation in contrast to feeling just tired based on their usual way of life in recent times. Each item (or situation such as sitting and reading) is rated on a 4-point Likert scale that ranges from "0 = Would never doze" to "3 = High chance of dozing." The total score on the Scale is the sum of the responses to each of the 8 items; therefore, the range of possible scores for each responder is 0 to 24. A total score of <10 indicates that the patient is not suffering from excessive daytime sleepiness. Individual items are not analyzed and have no independent, valid interpretations.

Subjects will complete the ESS at Screening.

#### 6 STATISTICAL ANALYSES

All programming and analyses will be performed using SAS software v9.4.

#### 6.1 STATISTICAL METHODOLOGY

#### 6.1.1 DETERMINATION OF SAMPLE SIZE

This study is designed to test non-inferiority (NI) of tolperisone doses relative to placebo, with a cyclobenzaprine test versus placebo to confirm the sensitivity of the simulator to detect treatment effects. The following assumptions were made in the sample size computation: (a) within-subject standard deviation for SDLP is approximately 6 cm; (b) the true difference between tolperisone doses and placebo is 0; and, (c) the NI margin is proposed to be 4.4 cm, which is the effect seen with 0.05% of blood alcohol content (BAC) with this driving simulator scenario. Under these assumptions, a sample of 30 subjects would provide in excess of 90% power to establish NI of tolperisone compared to placebo on any given dosing day in terms of the primary end point, SDLP. This sample size is considered more than adequate to detect cyclobenzaprine differences from placebo, which are anticipated to exceed the NI margin.

#### 6.1.2 ANALYSIS POPULATIONS

#### 6.1.2.1 SAFETY POPULATION

The Safety Population includes all subjects who received at least 1 dose of study drug, according to the treatment received in any given treatment period.

#### 6.1.2.2 INTENT-TO-TREAT (ITT) POPULATION

The Intent-to-Treat (ITT) Population includes all randomized subjects who receive at least 1 dose of study drug, according to the planned treatment in a given treatment period. This is the analysis population for efficacy analysis. Subjects will (in general) be included in all analyses for which data are non-missing.

### 6.1.2.3 PHARMACOKINETIC (PK) POPULATION

The Pharmacokinetic (PK) Population includes all subjects with evaluable plasma concentration data.

#### 6.1.3 STATISTICAL ANALYSES – GENERAL CONSIDERATIONS

In general, categorical variables will be summarized by the count (N) and percentage of subjects (%). Continuous variables will be summarized by the number of non-missing observations (N), mean, standard deviation (SD), median, minimum, and maximum values.

Formal statistical tests (where performed) will be two-sided and testing at the alpha=0.05 level of significance.

All study data are to be displayed in the data listings.

#### 6.1.4 MULTIPLE COMPARISONS

There are a number of comparisons of interest from which conclusions with respect to the NI of tolperisone vs. placebo will result. Initially, the statistical significance of the cyclobenzaprine vs. placebo (p<0.05) comparison is necessary to validate the experiment as having the ability to detect effects (i.e., assay sensitivity).

Subsequently, the NI of tolperisone to placebo (for initial dose, next day residual, and steady-state dose comparisons) will result in a conclusion of NI of tolperisone relative to placebo. For NI conclusions, the alternative hypothesis (of NI) will be considered established if the upper 95% confidence limit for tolperisone vs placebo difference is less than the pre-specified NI margin of 4.4 cm.

Cyclobenzaprine comparisons to placebo are to assess assay sensitivity and no adjustment to alpha levels will be made for either the comparison of

cyclobenzaprine to placebo or tolperisone, or for secondary endpoints or analyses.

The sequence of testing to control for multiplicity associated with comparisons of tolperisone to placebo (to assess NI) on multiple days is Day 1 (single-dose), followed by Day 3 (steady-state), followed by Day 2 (residual effect). Tolperisone will be considered NI to placebo if prior comparisons (at time points in the sequence provided, above) also indicate NI.

#### 6.1.5 PROCEDURES FOR HANDLING MISSING DATA

Subjects who discontinue, will only contribute to the pair-wise comparisons for which they have data.

For subjects that have incomplete data within an assessment, data will be listed but not summarized and/or analyzed for that assessment.

#### 6.2 SCREENING AND BASELINE CHARACTERISTICS

Summary tables will be constructed for the following screening or baseline data: demographic characteristics of age, sex, ethnic origin, height, weight and BMI for the safety population (Table 14.1.3), reason for screen failures (Table 14.1.4), medical history (Table 14.1.7), prior medications (Table 14.3.8.1), laboratory examinations (Tables 14.3.3.1-14.3.5.2), vital signs (Tables 14.3.6.1-14.3.6.5.3), and physical examination abnormalities (Table 14.3.8.1).

Data listings will be provided for the following screening and baseline data: screen failures (Listing 16.2.2.3), inclusion/exclusion criteria (Listing 16.2.3.2.1), inclusion/exclusion criteria violations (Listing 16.2.3.2.2), characteristics of age, sex, race, ethnicity (Listing 16.2.4.1), substance use (Listing 16.2.4.2, medical history (Listing 16.2.4.3), simulator sickness questionnaire (Listing 16.2.4.4), ESS (Listing 16.2.4.5), pharmacokinetic sampling (Listing 16.2.5.2), driving simulator (Listings 16.2.6.1.1-16.2.6.1.X), AEs (Listing 16.2.7.1) laboratory collections (Listing 16.2.8.1-16.2.8.3, urine drug screen, alcohol screen, and pregnancy test (Listing 16.2.8.4), prior medication (Listing 16.2.8.6.1), physical examination (Listing 16.2.8.7), 12-lead ECG (Listings 16.2.8.8.1 and 16.2.8.8.2), and vital signs, height, weight, and BMI (Listing 16.2.8.9).

#### 6.3 SUBJECT DISPOSITION

The number of subjects in each study population group will be presented by sequence (Table 14.1.1). The number of subjects randomized, completing each visit, discontinuing at each visit, and completing the study will be presented by

sequence (Table 14.1.2). A listing for study populations will be presented by subject (Listing 16.2.2.1).

For subjects discontinuing, individual subject information will be listed (Listing 16.2.1 respectively).

An important protocol deviation listing will be provided by subject (Listing 16.2.2.2). Deviations will be summarized category of deviation (Table 14.1.6).

Subjects excluded from the pharmacodynamics analyses will be listed (Listing 16.2.3.1).

#### 6.4 STUDY MEDICATION ADMINISTRATION

Study drug administration data will be listed by subject (Listing 16.2.5.1). The number of days exposed for each of the three treatment populations will be summarized (Table 14.1.5).

#### 6.5 PHARMACODYNAMIC ANALYSES

#### 6.5.1 PRIMARY ANALYSIS

The primary endpoint, SDLP, will be analyzed using a mixed model repeated measures with fixed effects for sequence, period, and treatment, with repeated observations for subjects. An unstructured covariance structure and Kenward-Roger degrees of freedom will be used. In the event an unstructured covariance structure fails to converge, a variance components covariance structure will be assumed.

In addition to assessments of treatment effect, p-values for significance testing of period and sequence effects will be provided.

Pair-wise comparisons (hypothesis tests) of differences in least squares means, and 95% confidence intervals on differences will be provided (Table 14.2.1.1) for:

#### Initial dose effect

- 1. cyclobenzaprine versus placebo following Day 1 PM dose
- tolperisone versus placebo following Day 1 PM dose
- 3. tolperisone versus cyclobenzaprine following Day 1 PM dose

#### Next day residual dose effect

- 4. cyclobenzaprine versus placebo following Day 2 AM dose
- 5. tolperisone versus placebo following Day 2 AM dose
- 6. tolperisone versus cyclobenzaprine following Day 2 AM dose

#### Steady-state dose effect

- 7. cyclobenzaprine versus placebo following Day 3 AM dose
- 8. tolperisone versus placebo following Day 3 AM dose
- 9. tolperisone versus cyclobenzaprine following Day 3 AM dose

In addition, pair-wise within-subject differences in SDLP greater than 4.4 cm in absolute value (equal to the previously found difference between placebo and 0.05% Blood Alcohol Content (BAC) for the CRCDS) will be compared using McNemar's test. Pair-wise, within subject differences in SDLP will also be tested for symmetry about zero (Laska 2012) using the maximally selected McNemar test (Table 14.2.1.2.1-14.2.1.2.9).

Summary statistics for raw values and change from baseline will be provided (mean, SD, median, minimum, maximum) for SDLP for each time point and treatment group. Figures will be provided for the within subject difference scores by treatment and day as both a histogram and scatter plot.

Data listings for driving simulator data will be provided (Listing 16.2.6.1.1-16.2.6.1.X).

#### 6.5.2 SECONDARY ANALYSES

Secondary endpoints of VAS, SDC, and driving performance endpoints will be evaluated and presented similarly, however Lane Exceedance will be log transformed (more specifically ln(x+1)) prior to analyses.

Tables will be presented in the same format as the primary output:

- VAS for motivation (Table 14.2.2.1)
- VAS for self-appraisal of driving performance (Table 14.2.2.2)
- Symbol Digit Coding:
  - Number of correct responses (Table 14.2.3.1)
  - Accuracy (Table 14.2.3.2)
  - Standard deviation of reaction time (Table 14.2.3.3)
- Other Driving Performance Endpoints
  - Lane exceedance; including number, maximum, and duration (Tables 14.2.4.1-14.2.4.3)
  - Average speed, speed deviation, excessive speeding count, speeding ratio (Tables 14.2.5.1-14.2.5.4)
  - Excessive Ay and Total Collisions(cornering speed threshold exceeded) (Table 14.2.6)

- Divided Attention (DA): Correct Responses, Omission Errors,
   Commission Errors, Reaction Time, Standard Deviation of Reaction
   Time (Tables 14.2.8.1-14.2.8.5)
- KSS (Table 14.2.9)

A data listing for KSS will be provided (Listing 16.2.6.2). A data listing for SDC will be provided (Listing 16.2.6.3). A data listing for the two VAS results will be provided (Listing 16.2.6.4).

### **Additional Secondary Analyses:**

#### **Total Collisions:**

Summary statistics will be provided (mean, SD, median, minimum, maximum) for total number of collisions for each time point and treatment group (Table 14.2.7). Additionally, differences in number of collisions for each pair-wise comparison will be provided with their corresponding Wilcoxon Signed Rank p-value. A bar chart will be provided pooling total number of collisions by 0, 1, 2, or >=3 for all 3 treatment groups.

### Self-reported readiness

Pair-wise comparisons for readiness to drive will be analyzed using McNemar's test (Table 14.2.10).

#### Plasma drug levels

Blood samples for the determination of plasma tolperisone concentrations will be drawn prior to each AM dosing on Days 1-3 and post-driving test (15-30 minutes after the drive) on Days 1 and 3. The relationship between initial dose effect, next day residual dose effect, and steady-state dose effect plasma drug levels and driving performance (i.e. the primary endpoint of SDLP) will be assessed by correlation. Both the Spearman and Pearson correlations will be reported (Tables 14.2.11.2-14.2.11.22).

#### 6.6 SAFETY ANALYSES

Safety analysis will be based on the safety population. Safety measures will be summarized using descriptive statistics and listed for each subject.

MedDRA thesaurus will be used to map AEs verbatim to preferred terms and body systems. WHOdrug thesaurus (Sep 1, 2016) will be used to map prior medication and concomitant medication verbatim to preferred terms and ATC Class.

#### 6.6.1 ADVERSE EVENTS (AE)

AEs will be coded using the Medical Dictionary for Regulatory Affairs (MedDRA version 20.0) coding system. Frequency tables will be presented by dose group summarizing:

- all treatment emergent AEs (Table 14.3.1.1),
- all treatment emergent treatment-related (defined as possibly or definitely related) AEs (Table 14.3.1.2),
- all serious treatment emergent AEs (Table 14.3.2.1)
- all AEs leading to discontinuation (Table 14.3.2.2).

Listings will be presented to provide:

- all AEs (Listing 16.2.7.1)
- all treatment related AEs (terms including definitely and probably related) (Listing 16.2.7.2).

#### 6.6.2 CLINICAL LABORATORY EVALUATIONS

Each laboratory examination observed value and change from baseline (when appropriate) will be summarized for hematology, blood chemistry, and urinalysis for each treatment at screening and end of study (Tables 14.3.2.1, 14.3.3.1, and 14.3.4.1). Shift tables will be constructed for hematology, blood chemistry, and urinalysis (Tables 14.3.2.2, 14.3.3.2, and 14.3.4.2).

Subject laboratory examination data listings will be provided (Listings 16.2.8.1-16.2.8.4). All clinical laboratory values outside normal range (including Screening/Visit 1 and EOS/Day 17 examination) will be listed by treatment and subject number, including demographic information and flagging of values (Listing 16.2.8.5).

#### 6.6.3 PHYSICAL EXAMINATION

A listing of physical examination data will be provided by subject (Listing 16.2.8.7.1). Subjects with any changes in the physical examination evaluation from Screening/Visit 1 to EOS/Day 17 will be listed (Listing 16.2.8.7.2).

#### 6.6.4 VITAL SIGNS

Summary statistics (n, mean, standard deviation, minimum, median, and maximum) will be presented for the raw values and change from baseline (defined as pre-dose Day 1 Period 1) values at each time point for all vital signs (including orthostatic vital signs) (Tables 14.3.6.1-14.3.6.5.3).

A data listing of vital sign data will be provided by treatment and subject (Listing 16.2.8.9).

#### 6.6.5 12-LEAD ELECTROCARDIOGRAM

Each ECG parameter observed value and change from screening will be summarized (Table 14.3.7.1). The ECG results will be categorized as normal, clinically significant abnormal, and not clinically significant abnormal. A shift table for ECG abnormalities will be provided (Table 14.3.7.2).

A data listing of ECG results for each parameter will be provided by subject (Listing 16.2.8.8.1). A data listing of ECG normality will be provided by subject (Listing 16.2.8.8.2).

#### 6.7 CONCOMITANT MEDICATIONS

Concomitant medications will be summarized (n and %) by ATC class and preferred term (Table 14.3.8.2).

Concomitant medications will be listed by subject (Listing 16.2.8.6.2).

#### 6.8 CONCENTRATION DATA

Concentration data will be summarized (n and %) by treatment (Table 14.2.11).

Concentration data will be listed by treatment and subject (Listing 16.2.5.2).

#### 6.9 ADDITIONAL COLLECTED DATA

General comments will be listed by subject (Listing 16.2.8.10).

#### 7 REFERENCES

Akerstedt T, Gillberg M. (1990). Subjective and objective sleepiness in the active individual. International Journal of Neuroscience, 52, 29–37.

CRCDS Operations Manual. Cognitive Research Corporation. Data on file.

Kaida M, Takahashi T, Åkerstedt A, Nakata Y, Otsuka T, Haratani K, et al. (2006). Validation of the Karolinska sleepiness scale against performance and EEG variables. Clinical Neurophysiology, 117, 1574–81.

Laska E, Meisner M, Wanderling J. A maximally selected test of symmetry about zero. Stat Med 2012;31:3178-91.

Siemen A, Gargano C, Cha J, Drexel M, Bautmans A, Heirman I, Laethem T, Hochadel T, Gheyle L, Bleys K, Beals C, Stoch A, Kay G, & Struyk A. (2015). A randomized, crossover, placebo-controlled clinical trial to assess the sensitivity of the CRCDS Mini-Sim to the next-day residual effects of zopiclone. Therapeutic Advances in Drug Safety, 6 (3), 86-97.

Wechsler, D. (1981). Wechsler Adult Intelligence Scale-Revised. San Antonio: Psychological Corporation.

## 8 TABLES, LISTINGS, AND FIGURES

Tables, listings, and figures numbering and titles will be finalized by the Sponsor at a later date.

#### 8.1 TABLES

| Table 14.1.1 | Study Populations |
|---|---|
| Table 14.1.2 | Subject Disposition (Safety population) |
| Table 14.1.3 | Subject Demographics (Safety population) |
| Table 14.1.4 | Reason for Screening Failures |
| Table 14.1.5 | Drug Exposure (Safety population) |
| Table 14.1.6 | Protocol Deviations (Safety population) |
| Table 14.1.7 | Medical History (Safety population) |
| Table 14.2.1.1 | Standard Deviation of Lateral Position (SDLP) (ITT Population) |
| Table 14.2.1.2.1 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Cyclobenzaprine versus Placebo Day 1 PM Dose) |
| Table 14.2.1.2.2 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Placebo Day 1 PM Dose) |
| Table 14.2.1.2.3 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Cyclobenzaprine Day 1 PM Dose) |
| Table 14.2.1.2.4 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Cyclobenzaprine versus Placebo Day 2 AM Dose) |
| Table 14.2.1.2.5 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Placebo Day 2 AM Dose) |
| Table 14.2.1.2.6 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Cyclobenzaprine Day 2 AM Dose) |
| Table 14.2.1.2.7 | Standard Deviation of Lateral Position (SDLP) Analysis of |

Breckenridge Statistics, Inc.: Statistical Analysis Plan-Neurana 115 Draft Version 1.0

| | Symmetry about Zero (ITT Population – Cyclobenzaprine versus Placebo Day 3 AM Dose) |
|---|---|
| Table 14.2.1.2.8 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Placebo Day 3 AM Dose) |
| Table 14.2.1.2.9 | Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population – Tolperisone versus Cyclobenzaprine Day 3 AM Dose) |
| Table 14.2.2.1 | Visual Analog Scale (VAS) Motivation (ITT Population) |
| Table 14.2.2.2 | Visual Analog Scale (VAS) Self-appraisal (ITT Population) |
| Table 14.2.3.1 | Symbol Digit coding (SDC) Number of Correct Responses (ITT Population) |
| Table 14.2.3.2 | Symbol Digit coding (SDC) Accuracy (ITT Population) |
| Table 14.2.3.3 | Symbol Digit coding (SDC) Standard Deviation of Reaction Time (ITT Population) |
| Table 14.2.4.1 | Driving Performance Lane Exceedance: Number (ITT Population) |
| Table 14.2.4.2 | Driving Performance Lane Exceedance: Maximum (ITT Population) |
| Table 14.2.4.3 | Driving Performance Lane Exceedance: Duration (ITT Population) |
| Table 14.2.5.1 | Driving Performance Average Speed (ITT Population) |
| Table 14.2.5.2 | Driving Performance Speed Deviation (ITT Population) |
| Table 14.2.5.3 | Driving Performance Excessive Speed Count (ITT Population) |
| Table 14.2.5.4 | Driving Performance Speeding Ratio (ITT Population) |
| Table 14.2.6 | Driving Performance Excessive Ay and Total Collisions (Cornering Speed Threshold Exceeded) (ITT Population) |
| Table 14.2.7 | Driving Performance Total Collisions (ITT Population) |
| Table 14.2.8.1 | Driving Performance Divided Attention – Correct Responses (ITT Population) |
| Table 14.2.8.2 | Driving Performance Divided Attention – Omission Errors (ITT Population) |
| Table 14.2.8.3 | Driving Performance Divided Attention – Commission Errors (ITT Population) |
| Table 14.2.8.4 | Driving Performance Divided Attention – Reaction Time (ITT Population) |
| Table 14.2.8.5 | Driving Performance Divided Attention – Standard Deviation of Reaction Time (ITT Population) |
| Table 14.2.9 | Karolinska Sleepiness Scale (KSS) (ITT Population) |
| Table 14.2.10 | Self-Reported Readiness (ITT Population) |

| Table 14.2.11.1 | Plasma Concentration by Time Point (Safety Population) |
|---|---|
| Table 14.2.11.2 | Correlation of In(Plasma Drug Levels) to SDLP |
| Table 14.2.11.3 | Correlation of In(Plasma Drug Levels) to Visual Analog Scale (VAS) Motivation |
| Table 14.2.11.4 | Correlation of In(Plasma Drug Levels) to Visual Analog Scale (VAS) Self-appraisal |
| Table 14.2.11.5 | Correlation of In(Plasma Drug Levels) to Symbol Digit Coding (SDC) Number of Correct Responses |
| Table 14.2.11.6 | Correlation of In(Plasma Drug Levels) to Symbol Digit Coding (SDC) Accuracy |
| Table 14.2.11.7 | Correlation of In(Plasma Drug Levels) to Symbol Digit Coding (SDC) Standard Deviation of Reaction Time |
| Table 14.2.11.8 | Correlation of In(Plasma Drug Levels) to Driving Performance Lane Exceedance Number |
| Table 14.2.11.9 | Correlation of In(Plasma Drug Levels) to Driving Performance Lane Exceedance Maximum |
| Table 14.2.11.10 | Correlation of In(Plasma Drug Levels) to Driving Performance Lane Exceedance Duration |
| Table 14.2.11.11 | Correlation of In(Plasma Drug Levels) to Driving Performance Average Speed |
| Table 14.2.11.12 | Correlation of In(Plasma Drug Levels) to Driving Performance Speed Deviation |
| Table 14.2.11.13 | Correlation of In(Plasma Drug Levels) to Driving Performance Speed Count |
| Table 14.2.11.14 | Correlation of In(Plasma Drug Levels) to Driving Performance Speeding Ratio |
| Table 14.2.11.15 | Correlation of In(Plasma Drug Levels) to Driving Performance Excessive Ay (Cornering Speed Threshold Exceeded) |
| Table 14.2.11.16 | Correlation of In(Plasma Drug Levels) to Driving Performance Total Collisions |
| Table 14.2.11.17 | Correlation of In(Plasma Drug Levels) to Driving Performance Divided Attention – Correct Responses |
| Table 14.2.11.18 | Correlation of In(Plasma Drug Levels) to Driving Performance Divided Attention – Omission Errors |
| Table 14.2.11.19 | Correlation of In(Plasma Drug Levels) to Driving Performance Divided Attention – Commission Errors |
| Table 14.2.11.20 | Correlation of In(Plasma Drug Levels) to Driving Performance Divided Attention – Reaction Time |
| Table 14.2.11.21 | Correlation of In(Plasma Drug Levels) to Driving Performance Divided Attention – Standard Deviation of Reaction Time |
| Table 14.2.11.22 | Correlation of In(Plasma Drug Levels) to Karolinska |

| | Sleepiness Scale (KSS) Pre-Drive |
|---|---|
| Table 14.3.1.1 | Treatment-Emergent Adverse Events by Maximum Severity (Safety Population) |
| Table 14.3.1.2 | Treatment-related, treatment-emergent adverse events by maximum severity (Safety Population) |
| Table 14.3.2.1 | Serious Adverse Events (Safety Population) |
| Table 14.3.2.2 | Adverse Events Leading to Discontinuation (Safety Population) |
| Table 14.3.3.1 | Hematology Change From Screening (Safety Population) |
| Table 14.3.3.2 | Hematology Shift Table (Safety Population) |
| Table 14.3.4.1 | Blood Chemistry Change From Screening (Safety Population) |
| Table 14.3.4.2 | Blood Chemistry Shift Table (Safety Population) |
| Table 14.3.5.1 | Urinalysis Change From Screening (Safety Population) |
| Table 14.3.5.2 | Urinalysis Shift Table (Safety Population) |
| Table 14.3.6.1 | Vital Sign Change from Baseline – Temperature (Safety population) |
| Table 14.3.6.2 | Vital Sign Change from Baseline – Respiration Rate (Safety population) |
| Table 14.3.6.3.1 | Vital Sign Change from Baseline – Supine Heart Rate (Safety population) |
| Table 14.3.6.3.2 | Vital Sign Change from Baseline – Standing Heart Rate (Safety population) |
| Table 14.3.6.3.3 | Vital Sign Change from Baseline – Orthostatic Heart Rate (Safety population) |
| Table 14.3.6.4.1 | Vital Sign Change from Baseline – Supine Systolic Blood Pressure (Safety population) |
| Table 14.3.6.4.2 | Vital Sign Change from Baseline – Standing Systolic Blood Pressure (Safety population) |
| Table 14.3.6.4.3 | Vital Sign Change from Baseline – Orthostatic Systolic Blood Pressure (Safety population) |
| Table 14.3.6.5.1 | Vital Sign Change from Baseline – Supine Diastolic Blood Pressure (Safety population) |
| Table 14.3.6.5.2 | Vital Sign Change from Baseline – Standing Diastolic Blood Pressure (Safety population) |
| Table 14.3.6.5.3 | Vital Sign Change from Baseline – Orthostatic Diastolic<br>Blood Pressure (Safety population) |
| Table 14.3.7.1 | ECG Change From Baseline (Safety population) |

| Table 14.3.7.2 | ECG Shift Table (Safety population) |
|----------------|---------------------------------------------|
| Table 14.3.8.1 | Prior Medication (Safety population) |
| Table 14.3.8.2 | Concomitant Medications (Safety population) |

## 8.2 LISTINGS

| Listing 16.2.1 | Subject Disposition (Safety Population) |
|---|---|
| Listing 16.2.2.1 | Study Population (Safety Population) |
| Listing 16.2.2.2 | Important Protocol Deviations (Safety Population) |
| Listing 16.2.2.3 | Screen Failures |
| Listing 16.2.3.1 | Subjects Who Were Excluded From ITT Population (Safety |
| | Population) |
| Listing 16.2.3.2.1 | Inclusion, Exclusion, and Eligibility Criteria Legend |
| Listing 16.2.3.2.2 | Inclusion and Exclusion Criteria Violations (Safety Population) |
| Listing 16.2.4.1 | Demographics and Baseline Characteristics (Safety Population) |
| Listing 16.2.4.2 | Substance Use (Safety Population) |
| Listing 16.2.4.3 | Medical History (Safety Population) |
| Listing 16.2.4.4 | Simulator Sickness Questionnaire (Safety Population) |
| Listing 16.2.4.5 | Epworth Sleepiness Scale (ESS) (Safety Population) |
| Listing 16.2.5.1 | Study Drug Administration (Safety Population) |
| Listing 16.2.5.2 | Plasma Concentration (Safety Population) |
| Listing 16.2.6.1.1 | Driving Simulator Part 1 of X (Safety Population) |
| Listing 16.2.6.1.X | Driving Simulator Part X of X (Safety Population) |
| Listing 16.2.6.2 | Karolinska Sleepiness Scale (KSS) (Safety Population) |
| Listing 16.2.6.3 | Cogscreen Symbol Digit Coding (SDC) (Safety Population) |
| Listing 16.2.6.4 | Visual Analog Scale (VAS) (Safety Population) |
| Listing 16.2.7.1 | Treatment-Emergent Adverse Events (Safety Population) |
| Listing 16.2.7.2 | Treatment-Related Treatment-Emergent Adverse Events (Safety Population) |
| Listing 16.2.8.1 | Hematology - Laboratory Collections (Safety Population) |
| Listing 16.2.8.2 | Blood Chemistry - Laboratory Collections (Safety Population) |
| Listing 16.2.8.3 | Urinalysis - Laboratory Collections (Safety Population) |
| Listing 16.2.8.4 | Drug Screen, Alcohol Screen, Pregnancy, HCV-AB, HbsAg, HIV |
| | Test Results (Safety Population) |
| Listing 16.2.8.5 | Laboratory Values Outside of Normal Range (Safety Population) |
| Listing 16.2.8.6.1 | Prior Medications (Safety Population) |
| Listing 16.2.8.6.2 | Concomitant Medications (Safety Population) |

Breckenridge Statistics, Inc.: Statistical Analysis Plan-Neurana 115 Draft Version 1.0

| Listing 16.2.8.7.1 | Physical Examination (Safety Population) |
|---|---|
| Listing 16.2.8.7.2 | Shift in Physical Examination (Safety Population) |
| Listing 16.2.8.8.1 | 12-Lead Electrocardiogram Results (Safety Population) |
| Listing 16.2.8.8.2 | 12-Lead Electrocardiogram Assessment (Safety Population) |
| Listing 16.2.8.9 | Vital Signs (Safety Population) |
| Listing 16.2.8.10 | General Comments (Safety Population) |

### 8.3 FIGURES

| F: 440444 | M |
|---|---|
| Figure 14.2.1.1.1 | Within Subject Difference Scores in SDLP by Treatment |
| Figure 14.2.1.2.1 | Within Subject Difference Scores (Cyclobenzaprine - Placebo) |
| 1 iguic 14.2.1.2.1 | (ITT Population - Day 1 PM Dose) |
| Figure 14 2 1 2 2 | Within Subject Difference Scores (Tolperisone - Placebo) (ITT |
| Figure 14.2.1.2.2 | Population – Day 1 PM Dose) |
| Figure 14 0 1 0 2 | Within Subject Difference Scores (Tolperisone - |
| Figure 14.2.1.2.3 | Cyclobenzaprine) (ITT Population – Day 1 PM Dose) |
| F: 440404 | Within Subject Difference Scores (Cyclobenzaprine - Placebo) |
| Figure 14.2.1.2.4 | (ITT Population - Day 2 AM Dose) |
| F: 44 0 4 0 5 | Within Subject Difference Scores (Tolperisone - Placebo) (ITT |
| Figure 14.2.1.2.5 | Population – Day 2 AM Dose) |
| F: 44 0 4 0 C | Within Subject Difference Scores (Tolperisone - |
| Figure 14.2.1.2.6 | Cyclobenzaprine) (ITT Population – Day 2 AM Dose) |
| F: 440407 | Within Subject Difference Scores (Cyclobenzaprine - Placebo) |
| Figure 14.2.1.2.7 | (ITT Population - Day 3 AM Dose) |
| F: 44 0 4 0 0 | Within Subject Difference Scores (Tolperisone - Placebo) (ITT |
| Figure 14.2.1.2.8 | Population – Day 3 AM Dose) |
| F: 440400 | Within Subject Difference Scores (Tolperisone - |
| Figure 14.2.1.2.9 | Cyclobenzaprine) (ITT Population – Day 3 AM Dose) |
| F: 4404404 | Within Subject Difference Scores in SDLP by Plasma |
| Figure 14.2.11.2.1 | Concentration for Tolperisone Day 1 |
| Fig 44 0 44 0 0 | Within Subject Difference Scores in SDLP by Plasma |
| Figure 14.2.11.2.2 | Concentration for Tolperisone Day 2 |
| Fig. 44 0 44 0 0 | Within Subject Difference Scores in SDLP by Plasma |
| Figure 14.2.11.2.3 | Concentration for Tolperisone Day 3 |
| Figure 14.2.7 | Total Collisions |
| | 1 |

#### Neurana Pharmaceuticals Inc.


Neurana 115
Page X of Y

Neurana 115
Table 14.1.1

Table 14.1.1 Study Populations

| | Placebo | Tolperisone 450 mg | Cyclobenzaprine 30 mg | Overall |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Study Population | n (%) | n (%) | n (%) | n (%) |
| Screening Failures | | | | XX |
| Safety Population* | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| ITT Population** | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| per p. 3 of the delay | | | | |

PK Population \*\*\*

<sup>\*</sup> The Safety Population includes all subjects who received at least 1 dose of study drug

<sup>\*\*</sup> The Intent-to-Treat (ITT) Population includes all randomized subjects who receive at least 1 dose of study drug in a given treatment period. This is the analysis population for efficacy analysis. Subjects will (in general) be included in all analyses for which data are non-missing.

<sup>\*\*\*</sup> The Pharmacokinetic (PK) Population includes all subjects with evaluable plasma concentration data. SAS Program Name: Date: Source Data: Listing 16.2.2.1

#### Neurana Pharmaceuticals Inc.


Neurana 115

Table 14.1.2 Subject Disposition (Safety Population)

| | | Placebo | | Tolperisone<br>450 mg | | Cyclobenzaprine<br>30 mg | | Overall | |
|---|---|---|---|---|---|---|---|---|---|
| Study Population | | , | (%) | , | (%) | • | =xx)<br>(%) | • | (%) |
| Completed Study | | XX | XX.X | XX | xx.x | XX | xx.x | xx | XX.X |
| Withdrew From Study | | xx | XX.X | XX | xx.x | XX | xx.x | XX | xx.x |
| XXXXXXX | | xx | XX.X | XX | xx.x | XX | xx.x | XX | XX.X |
| ҮҮҮҮҮҮҮ | | XX | XX.X | XX | XX.X | XX | XX.X | xx | XX.X |
| SAS Program Name: | Date: | | | | Sour | rce Data: | Listing | g 16.2 | .2.1 |


Neurana 115
Page X of Y

Neurana 115

Table 14.1.3
Demographics and Baseline Characteristics (Safety Population)

| | | | P] | Lacebo | Tolper | risone 450<br>mg | | oenzaprine<br>30 mg | 70 | verall |
|---|---|---|---|---|---|---|---|---|---|---|
| Characteristic | | ( | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | |
| Age | | | | | | | | | | |
| N | | | | XX | | xx | | xx | | xx |
| Mean (SD) | | | XX.X | (xx.xx) | XX.X | (xx.xx) | XX.X | (xx.xx) | xx.x | (xx.xx) |
| Median | | | | XX.X | | XX.X | | XX.X | | XX.X |
| Minimum, Maxi | muı | m | XX.X | , xx.x | XX.X | xx.x , xx.x | | XX.X , XX.X | | xx.x , xx.x |
| Sex | | | XX | (xx.x) | XX | (xx.x) | xx | (xx.x) | XX | (xx.x) |
| Male | n | (왕) | XX | (xx.x) | xx | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Female | n | (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Race | | | | | | | | | | |
| Caucasian | n | (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Black | n | (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Hispanic | n | (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Asian | n | (왕) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Native American | n | (왕) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Other | n | (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Ethnicity | | | | | | | | | | |
| Hispanic or | | | | , , | | , , | | | | , |
| Latino<br>Not Hispanic or | n | (응) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Latino | n | (%) | XX | (xx.x) | xx | (xx.x) | xx | (xx.x) | XX | (xx.x) |
| Height (cm) | | | | | | | | | | |
| N | | | | XX | | xx | | xx | | XX |
| Mean (SD) | | | XX.X | (xx.xx) | XX.X | (xx.xx) | XX.X | (xx.xx) | xx.x | (xx.xx) |
| Median | | | | XX.X | | XX.X | | XX.X | | xx.x |
| Minimum, Maxi | mui | m | XX.X | , xx.x | XX.X | , xx.x | XX.X | x , xx.x | XX. | , xx.x |
| Weight (kg) | | | | | | | | | | |

| Mourana | Pharmacei | iticala | Inc |
|---------|-----------|---------|-----|
| neurana | Pharmacei | ulicais | mc. |


| | N | XX | XX | XX | xx |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Minimum, Maximum | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |
| BMI | (kg/m^2) | | | | |
| | N | XX | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median xx.x | | XX.X | XX.X | xx.x |
| | Minimum, Maximum | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |

SAS Program Name:

Date:

Source Data: Listing 16.2.4.1 and Listing 16.2.8.9

Neurana 115

Table 14.1.4
Reason for Screening Failures

Overall

| | (N | =xx) |
|-----------|----|------|
| | n | (응) |
| Reason #1 | xx | XX.X |
| etc | xx | XX.X |
| | XX | XX.X |
| | XX | XX.X |
| | XX | xx.x |
| | XX | XX.X |
| | XX | XX.X |
| | XX | XX.X |
| | XX | XX.X |
| | XX | xx.x |

Source Data: Listing 16.2.2.3

Neurana 115
Page X of Y

Neurana 115

Table 14.1.5
Drug Exposure
(Safety Population)

Source Data: Listing 16.2.5.1

| | Placebo | Tolperisone 450<br>mg | Cyclobenzaprine<br>30 mg | Overall |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Days | | | | |
| N | XX | XX | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX.X , XX.X | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |

| Neurana Pharmaceuticals Inc | Neurana | Pharmaceu | uticals | Inc. |
|-----------------------------|---------|-----------|---------|------|
|-----------------------------|---------|-----------|---------|------|

Neurana 115
Page X of Y

Neurana 115

Table 14.1.6
Protocol Deviations
(Safety Population)

| | Overall<br>(N=xx) |
|--------------------|-------------------|
| Deviation Category | n (%) |
| xxxx | xx (xx.xx) |
| УУУУ | xx (xx.xx) |

SAS Program Name:

Date:

Source Data: Listing 16.2.2.2


Neurana 115

Table 14.1.7 Medical History (Safety Population)

Overall

| | (N=xx) |
|----------|-----------|
| Category | n % |
| HEENT | xx (xx.x) |
| etc | xx (xx.x) |

Subjects with more than one occurrence in a category are only counted once.

SAS Program Name:

Date: Source Data: Listing 16.2.4.3


Neurana 115 Page x of y

Table 14.2.1.1
Standard Deviation of Lateral Position (SDLP)
(ITT Population)

| | | | | Cyclobenzaprine 30 | |
|---|---|---|---|---|---|
| | | Placebo | Tolperisone 450 mg | mg | |
| Day | | (N=xx) | (N=xx) | (N=xx) | |
| Day X | N | XX | xx | xx | |
| | Mean (SD) | xx.xxxx (xx.xx) | xx.xxxx (xx.xx) | xx.xxxx (xx.xx) | |
| | Median | XX.X | XX.X | XX.X | |
| | Min, Max | xx.xxxx , xx.xxxx | xx.xxxx , xx.xxxx | xx.xxxx , xx.xxxx | |
| | | Model Fixed Effects of Interest | Tolperisone 450 mg<br>vs PBO | Cyclobenzaprine vs<br>PBO | Tolperisone 450 mg vs Cyclobenzaprine |
| | Diff in LSMean | | XX.XXXX | XX.XXXX | xx.xxx |
| | 95%CI* | | (xx.xx, xx.xx) | (xx.xx , xx.xx) | (xx.xx, xx.xx) |
| | p-value Treatment* | | 0.xxxx | 0.xxxx | 0.xxxx |
| | p-value Sequence* | 0.xxxx | | | |
| | p-value Period* | 0.xxxx | | | |

Repeat table for VAS, SDC, KSS, and other driving performance measures (see SAP for proposed table list). Mixed model repeated measures with fixed effects for sequence, period, and treatment, repeated assessments for subjects, unstructured covariance structure, and Kenward-Roger degrees of freedom.

SAS Program Name:

Date:

Source Data: Listing 16.2.6.1.X


Page 10 Neurana 11<u>5</u>

Neurana 115 Page x of y

Table 14.2.1.2.1

Standard Deviation of Lateral Position (SDLP) Analysis of Symmetry about Zero (ITT Population - Cyclobenzaprine 30 mg versus Placebo)

| Threshold | Sign | Low | Neutral | High | McNemar | Nominal P-value |
|-----------|------|-----|---------|------|---------|-----------------|
| x.xxx | -/+ | XX | xx | xx | x.xxxx | 0.xxxxx |
| x.xxxx | -/+ | xx | XX | xx | x.xxxx | 0.xxxxx |

Repeat for each comparison

SAS Program Name: Date: Source Data: Listing 16.2.6.1.X


Neurana 115

Page x of y

Table 14.2.7
Driving Performance Total Collisions
(ITT Population)

| | | Placebo | Tolperisone 450<br>mg | Cyclobenzaprine<br>30 mg | |
|---|---|---|---|---|---|
| Day | Statistic | (N=xx) | (N=xx) | (N=xx) | |
| Day 1 | N | XX | XX | XX | |
| | Mean | X . X | X.X | X • X | |
| | SD | X.XX | x.xx | X.XX | |
| | Median | X . X | X.X | X • X | |
| | Min, Max | xx, xx | xx, xx | xx, xx | |
| | Diff in # of Coll | isions | Tolperisone 450<br>vs PBO | Cyclobenzaprine<br>30 mg | Tolperisone vs<br>Cyclobenzaprine |
| | N | | XX | XX | XX |
| | Mean | | X • X | X.X | X . X |
| | SD | | X.XX | X.XX | X.XX |
| | Median | | X • X | X.X | X.X |
| | Min, Max | | xx, xx | XX, XX | XX, XX |
| etc | p-value* | | 0.xxxx | 0.xxxx | 0.xxxx |

### \*Wilcoxon Signed Ranks test.

SAS Program Name: Date: Source Data: Listing 16.2.6.1.X


Neurana 115

Table 14.2.12 Self-Reported Readiness (ITT Population)

| | | First Treatment | Second Treatment | N(%) | |
|---|---|---|---|---|---|
| Day | Comparison | | | | p-value* |
| Day 1 | xxxxxxxxxxxx | No | No | xx (xxx.x%) | 0.xxxx |
| | | Yes | No | xx (xxx.x%) | 0.xxxx |
| | | No | Yes | xx (xxx.x%) | 0.xxxx |
| | | Yes | Yes | xx (xxx.x%) | 0.xxxx |

\*McNemar's test.

SAS Program Name: Date: Source Data: Listing 16.2.6.X


Neurana 115 Page x of y

Table 14.2.11.1
Plasma Concentration
(PK Population)

Min, Max

SAS Program Name: Date: Source Data: Listing 16.2.5.2

xx.xxxx , xx.xxxx


Neurana 115 Page x of y

Table 14.2.11.2 Correlation of ln(Plasma Drug Levels) to SDLP (ITT Population)

Tolperisone 450 mg

Day X Pearson Correlation x.xxxx
Spearman Correlation x.xxxx

SAS Program Name: Date: Source Data: Listings 16.2.5.2 and 16.2.6.1.1

Neurana 115 Page X of Y

Table 14.3.1.1

Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity (Safety population)

| Primary System Organ Class\ Preferred Term\ | Placebo<br>(N=xx) | Tolperisone 450 mg (N=xx) | Cyclobenzaprine<br>30 mg<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Severity | n(%) | n(%) | n (%) | n(%) |
| Total Number of Adverse Events | XXX | XXX | XXX | XXX |
| Any primary system organ class | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Mild | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Moderate | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Severe | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| SOC 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Mild | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Moderate | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Severe | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Preferred Term 1 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Mild | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Moderate | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Severe | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Etc

NOTE FOR PROGRAMMING: repeat table for treatment related (with footnote defining related) 14.3.1.2

Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class alphabetically. Subjects with more than one occurrence in a category are only counted once.

SAS Program Name:

Date:

Source Data: Listing 16.2.7.1


Neurana 115
Page X of Y

Neurana 115 Page X

Table 14.3.2.1
Serious Adverse Events
(Safety Population)

Treatment:

| Subjec<br>No./ | | | AE Term/<br>Preferred | Start<br>Date/ | End | | | | Relationshi | - | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age/ | Subjec | t AE | Term/ | Start | Date/ | | Maximum | | to Study | Taken | | |
| Sex | No. | Seq Numbe | erSOC Class | Time | End Tir | neFrequency | Severity | Serious | s?Drug | Due to A | EOutcome | Sequelae |
| XX-XXX | xx-xxx | XXX XX | XXXXXXXXX | x YYYYMMI | DD YYYYMMI | DDSingle Episode/ | Mild/ | Yes | Unrelated/ | No | Resolved | XXXXXXXXX |
| XX | | | XXXXXXXXX | hh:mm | hh:mm | Intermittent/Continuo | usModerate | / | Possibly | Action/ | without | |
| /X | | | XXXXXXXXX | | | | Severe | | Related/ | etc | Sequelae/ | |
| | | | | | | | | | Definitely | | etc | |
| | | | | | | | | | Related | | | |

Repeat for AE leading to discontinuation Table 14.3.2.2 A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name:

Date:

NOTE TO PROGRAMMER: screening, placebo, 450 mg tolperisone, 30 mg cyclobenzaprine


Neurana 115 Page x of y

Table 14.3.3.1
Hematology Change From Screening
(Safety population)

| Labtest (Units) | | Overall (N=xx) |
|---|---|---|
| Screening | | |
| Observed | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.xxx (xx.xxx)<br>xx.xxx<br>xx.x , xx.x |
| End of Study<br>Observed | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.xxx (xx.xxx)<br>xx.xxx<br>xx.x , xx.x |
| End of Study<br>Change from<br>Screening | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.xxx (xx.xxx)<br>xx.xxx<br>xx.x , xx.x |

[repeat for each lab/parameter]

NOTE FOR PROGRAMMING: Repeat for blood chemistry (Table 14.3.4.1), urinalysis (Table 14.3.5.1), and ECG (Table 14.3.7.1)

Change N reflects number of subjects with both screening and end of study evaluation.

SAS Program Name: Date: Source Data: Listing 16.2.8.1


Neurana 115 Page x of y

Table 14.3.3.2 Hematology Shift Table (Safety Population)

Overall

Laboratory
Examination

Shift Category

n (%)

XXXXXXXXXX

LOW TO LOW

XX (XX.X)

LOW TO NORMAL

XX (XX.X)

[repeat for each lab]
NOTE FOR PROGRAMMING: Repeat for blood chemistry (Table 14.3.4.2), urinalysis (Table 14.3.5.2), and ECG (Table 14.3.7.2).

SAS Program Name: Date: Source Data: Listing 16.2.8.1


Neurana 115 Page X of Y

Table 14.3.6.3.1

Vital Signs Change From Baseline - Supine Heart Rate
(Safety population)

| Heart Rate (bpm) | | Overall (N=xx) | Placebo (N=xx) | Tolperisone<br>450 mg<br>(N=xx) | Cyclobenzaprine<br>30 mg<br>(N=xx) |
|---|---|---|---|---|---|
| Screening | | (11 1111) | | | _ |
| Observed | n | XX | | | |
| ODSELVEG | Mean (SD) | xx.x (xx.xx) | | | |
| | Min, Max | | | | |
| | MIII, Max | xx.x , xx.x | | | |
| Day 1 Pre-dose | | | | | |
| Observed | n | | XX | XX | xx |
| | Mean (SD) | | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Min, Max | | xx.x , xx.x | xx.x , xx.x | XX.X , XX.X |
| etc | | | | | |
| Observed | n | | XX | XX | xx |
| Observed | Mean (SD) | | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Min, Max | | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |
| etc | | | | | |
| Change | n | | xx | XX | xx |
| <u> </u> | Mean (SD) | | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Min, Max | | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |

[repeat for all post dose measurements]

NOTE FOR PROGRAMMING: Repeat for all vitals tables

Note for programming trt columns populated for visits after baseline visit. Orthostatic tables need footnote defining standing-supine.

Baseline defined as pre-dose Day 1.

Note: Change N reflects number of subjects with both baseline and at least one post-dose assessment.

SAS Program Name: Date: Source Data: Listing 16.2.8.9

[repeat for all ingredients and ATC

classes/ingredients]


Neurana 115

Table 14.3.8.1 Prior Medications (Safety population)

| | Overall |
|-------------------------------|---------|
| | (N=xx) |
| ATC Class/Preferred Term | n % |
| Any ATC Class with medication | xx xx.x |
| ATC Therapeutic Class 1 | |
| -Total | xx xx.x |
| Ingredient 1 | xx xx.x |
| Ingredient 2 | xx xx.x |
| Ingredient 3 | XX XX.X |
| ATC Therapeutic Class 2 | XX XX.X |
| -Total | XX XX.X |
| Ingredient 1 | XX XX.X |
| Ingredient 2 | XX XX.X |
| etc. | |

ATC classes are presented alphabetically; preferred terms are sorted within ATC class alphabetically. Subjects with more than one occurrence in a category are only counted once.

SAS Program Name:

Date:

Source Data: Listing 16.2.8.6.1

Neurana 115


Neurana 115
Page X of Y

Table 14.3.8.2 Concomitant Medications

Concomitant Medications (Safety population)

Overall

(N=xx)

| ATC Class/Preferred Term | 1 | n % |
|---------------------------------------|----|------|
| Any ATC Class with medication/surgery | XX | xx.x |
| ATC Therapeutic Class 1 | | |
| -Total | XX | xx.x |
| Ingredient 1 | XX | xx.x |
| Ingredient 2 | XX | xx.x |
| Ingredient 3 | XX | XX.X |
| ATC Therapeutic Class 2 | XX | XX.X |
| -Total | XX | XX.X |
| Ingredient 1 | XX | XX.X |
| Ingredient 2 | XX | XX.X |

etc.

[repeat for all ingredients and ATC
classes/ingredients]

ATC classes are presented alphabetically; preferred terms are sorted within ATC class alphabetically. Subjects with more than one occurrence in a category are only counted once.

SAS Program Name:

Date:

Source Data: Listing 16.2.8.6.2

| Neurana Pharmaceuticals Inc |
|-----------------------------|
|-----------------------------|


Neurana 115

Listing 16.2.1 Subject Disposition (Safety Population)

| Subject No. | Sequence | Visit<br>Date | Completed /<br>Premature<br>Withdrawal | Date | Reason for Withdrawal |
|---|---|---|---|---|---|
| xx-xxx | XXX | YYYYMMDD | Completed /<br>Withdrew | YYYYMMDD | Adverse Event<br>etc |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115
Page X of Y

Neurana 115

Listing 16.2.2.1 Study Population

| Subject No. | Sequence | Safety* | ITT** | PK*** |
|-------------|----------|---------|--------|--------|
| xx-xxx | XXX | Yes/no | Yes/no | Yes/no |
| xx-xxx | XXX | Yes/no | Yes/no | Yes/no |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine

SAS Program Name:

Date:

<sup>\*</sup> The Safety Population includes all subjects who received at least 1 dose of study drug

<sup>\*\*</sup> The Intent-to-Treat (ITT) Population includes all randomized subjects who receive at least 1 dose of study drug in a given treatment period. This is the analysis population for efficacy analysis. Subjects will (in general) be included in all analyses for which data are non-missing.

<sup>\*\*\*</sup> The Pharmacokinetic (PK) Population includes all subjects with evaluable plasma concentration data.


Neurana 115
Page X of Y

Neurana 115

Listing 16.2.2.2
Important Protocol Deviations
(Safety Population)

| Subject No. | Sequence | Deviation Category | Description of Deviation |
|-------------|----------|---------------------|--------------------------|
| XX-XXX | XXX | xxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxx |

| Maurana | Pharmacei | ıticəle | Inc |
|---------|-----------|---------|------|
| neurana | Fuaimacei | มแผลเธ | HIG. |

Neurana 115
Page X of Y

Neurana 115

Listing 16.2.2.3 Screen Failures

| | | | | | | | | | | Reason |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Date of | | | | | | for |
| Investigator | Screening | | | Informed | | | | Race | | Screen |
| No. | Number | Visit Date | Date of Birth | Consent | Age | Sex | Race | Other | Ethnicity | Failure |
| · | | | | | | | | | | |
| XX | XXX | YYYYMMDD | YYYYMMDD | YYYYMMDD | XXX | Female | XXXXXX | XXXXXXXX | XXXXXXXX | XXXXXXXX |

SAS Program Name:

Date:


Neurana 115 Page X of Y

Listing 16.2.3.1
Subjects Who Were Excluded From ITT Population (Safety Population)

#### Neurana Pharmaceuticals Inc. Confidential Page 6 Neurana 115 Page X of Y SAP Version Final 1.0

Neurana 115

Listing 16.2.3.2.1 Inclusion, Exclusion, and Eligibility Criteria Legend

To be populated


Neurana 115

Listing 16.2.3.2.2
Inclusion and Exclusion Criteria Violations (Safety Population)

| Subject<br>No. | Sequence | Visit | Category | Question<br>Number | Inclusion/Exclusion<br>Question | Result |
|---|---|---|---|---|---|---|
| xx-xxx | XXX | XXXX | XXXXXXXXX | XXXXXXX | XXXXXXXXXXXXXXX | X |


Neurana 115
Page X of Y

Neurana 115

Listing 16.2.4.1
Demographics and Baseline Characteristics
(Safety Population)

| Subject No. | Sequence | Visit<br>Date | Date of<br>Birth | Date of<br>Informed<br>Consent | Age | Sex | Race | Race Other | Ethnicity |
|---|---|---|---|---|---|---|---|---|---|
| xx-x | XXX | YYYYMMDD | YYYYMMDD | YYYYMMDD | xxx | Female | xxxxxx | xxxxxx | xxxxxxxxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.4.2
Substance Use
(Safety Population)

| Subject No. | Sequence | Status | Substance | Quantity | Frequency | Start Date | End Date |
|---|---|---|---|---|---|---|---|
| XX-XXX | XXX | XXXXXXXXXXXX | XX | XX | XX | YYYYMMDD | YYYYMMDD |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.4.3 Medical History (Safety Population)

| Subject No. | Sequence | Date of Visit | System | Condition | Date of<br>Diagnosis | Status | |
|---|---|---|---|---|---|---|---|
| xx-xxx | XXX | YYYYMMDD | xxxxxx | ****** | YYYYMMDD Resolved. | Stable. | Unstable |


Neurana 115

Listing 16.2.4.4 Simulator Sickness Questionnaire (Safety Population)

| Subject No. | Sequence | Date of Visit | Was the Simulator Sickness<br>Questionnaire Completed? |
|---|---|---|---|
| xx-xxx | XXX | YYYYMMDD | Yes/No |


Neurana 115

Listing 16.2.4.5
Epworth Sleepiness Scale (ESS)
(Safety Population)

| Subject No. | Sequence | Date of Visit | Situation | Result |
|-------------|----------|---------------|----------------|--------|
| xx-xxx | XXX | YYYYMMDD | xxxxxxxxxxxxxx | 0-3 |


Neurana 115

Listing 16.2.5.1
Study Drug Administration
(Safety Population)

Treatment:

| Subject | | Visit | | Date of | ${\tt Randomization}$ | Date of | Time of |
|---|---|---|---|---|---|---|---|
| Number | Sequence | Date | Visit | Randomization | Number | Administration | Administration |
| xx-xxx | XXX | YYYYMMDD | xxxxx | YYYYMMDD | xxx | YYYYMMDD | hh:mm |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:

NOTE TO PROGRAMMER: placebo, 450 mg tolperisone, 30 mg cyclobenzaprine


Neurana 115

Listing 16.2.5.2 Plasma Concentration (Safety Population)

Treatment:

| Subject | | | | | | Date of | Time of | |
|---|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit Date | Visit | Time Point | Not Done | Draw | Draw | Concentration |
| xx-xxx | XXX | YYYYMMDD | XXXXXXXX | XXXXX | XXXX | YYYYMMDD | hh:mm | XXXXX.XX |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine
SAS Program Name:

NOTE TO PROGRAMMER: placebo, 450 mg tolperisone, 30 mg cyclobenzaprine


Neurana 115

Listing 16.2.6.1.1
Driving Simulator Part 1 of X
(Safety Population)

Treatment:

| Subject | | | | Not | Start | Start | Feel Safe to | Columns |
|---|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit | Test | Done | Date | Time | Drive? | TBD |
| xx-xxx | XXX | xxxx x | ***** | xxx | YYYYMMDD | hh:mm | Yes/No | XX.XX |


Neurana 115

Listing 16.2.6.1.X
Driving Simulator Part X of X
(Safety Population)

Treatment:

| Subject | | | Visit | Feel | Safe | to | Columns |
|---------|-------------|------|----------|------|-------|----|---------|
| No. | Sequence V: | isit | Date | Dı | rive? | | TBD |
| xx-xxx | XXX x | XXX | YYYYMMDD | Υe | es/No | | XX.XX |


Neurana 115

Listing 16.2.6.2
Karolinska Sleepiness Scale (KSS)
(Safety Population)

Treatment:

| Subject<br>No. | Sequence | Visit | Visit Date | Test | Not Done | Start Date Start Time Score (1-9) |
|---|---|---|---|---|---|---|
| xx-xxx | xxx | xxxxxxx | YYYYMMDD | Pre-Dose/<br>Post-Dose | xxxx | YYYYMMDD hh:mm x |

NOTE TO PROGRAMMER: placebo, 450 mg tolperisone, 30 mg cyclobenzaprine

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.6.3
Cogscreen Symbol Digit Coding (SDC)
(Safety Population)

Treatment:

| xx-xxx | XXX | xxxxx | Yes/no | YYYYMMDD | XX.XX | xxxxxxxxx | XX | xxx.xx | x.xxx |
|---|---|---|---|---|---|---|---|---|---|
| No. | Sequence' | Visit | Done | Date | Time | Test | Responses | Accuracy | Variability |
| Subject | 5 | | Not | Start | Start | | Correct | | Speed |
| | | | | | | | Number of | | |
| | | | | | | | Total | | |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine

SAS Program Name: Date:

NOTE TO PROGRAMMER: placebo, 450 mg tolperisone, 30 mg cyclobenzaprine


Neurana 115

Listing 16.2.6.4

Self-Rating of Driving Simulator Performance Visual Analog Scale (VAS) (Safety Population)

| | XXX | xxxxxx | YYYYMMDD | Yes/blank | xxx | Yes/mm |
|---|---|---|---|---|---|---|
| NO. | | | Date | | The Last 60 Minutes? | Best During Your Last 60 Minutes of Driving? |
| NT | Sequence | Visit | Date | Not Done | mba Taat CO | Deat Dunian Valle Test |
| Subject | Sequence | | Visit | Not Done | Think You Drove For | Feel To Drive At Your |
| | | | | | How Well do You | How Motivated Did You |
#### Neurana Pharmaceuticals Inc. Confidential SAP Version Final 1.0

Neurana 115 Page X of Y Neurana 115

Listing 16.2.7.1 Adverse Events (Safety Population) Page 20

Treatment:

| Subject | 5 | | AE Term/ | Start | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No./ | | | Preferred | Date/ | End | | | | Relationshi | pAction | | |
| Age/ | Subject | : AE | Term/ | Start | Date/ | | Maximum | | to Study | Taken | | |
| Sex | No. | Seq Numbe | rSOC Class | Time | End Tim | eFrequency | Severity | Serious | ?Drug | Due to A | EOutcome | Sequelae |
| xx-xxx | / <sub>XX-XXX</sub> | XXX xx | XXXXXXXXX | x YYYYMMI | D YYYYMMD | DSingle Episode/ | Mild/ | Yes/no | Unrelated/ | No | Resolved | XXXXXXXXX |
| XX | | | XXXXXXXXX | hh:mm | hh:mm | Intermittent/Continuou | ısModerate | / | Possibly | Action/ | without | |
| /X | | | XXXXXXXXX | | | | Severe | | Related/ | etc | Sequelae/ | |
| | | | | | | | | | Definitely | | etc | |
| | | | | | | | | | Related | | | |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine Date:

#### Confidential SAP Version Final 1.0


Neurana 115

Listing 16.2.7.2

Treatment-Related, Treatment-Emergent Adverse Events (Safety Population)

#### Treatment:

| Subject<br>No./<br>Age/<br>Sex Seg | AE<br>Numbe | AE Term/ Preferred Term/ rSOC Class | Start<br>Date/<br>Start<br>Time | End<br>Date/<br>End Tim | eFreguency | Maximum<br>Severity | Serious: | to Study | pAction Taken<br>with Study<br>Medication | Action<br>Taken<br>to Treat<br>AE | Outcome | Seguelae |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sex Seq<br>xx-xxx/XXX<br>xx<br>/X | | r SOC Class xxxxxxxxxx xxxxxxxxx xxxxxxxxx | | | eFrequency<br>DSingle Episode/<br>Intermittent/Continuou | Severity<br>Mild/<br>sModerate/<br>Severe | Yes/no | PDrug<br>Unrelated/<br>Possibly<br>Related/<br>Probably<br>Related | None/ Dosage Increased/ Dose Reduced/ Dose Interrupted/ Dose | No Action/ Subject Withdrawn from Study/ Treatment Given/ Other | Resolved without Sequelae/ nResolved with Sequelae/ | Sequelae<br>xxxxxxxxxx |
| | | | | | | | | | applicable | | to Death/ Resolved with Death: Event did not Contribute to Death/ Ongoing/ Lost to Follow-Up | • |


Neurana 115

Listing 16.2.8.1
Hematology - Laboratory Collections
(Safety Population)

Treatment:

| Subject | | | Date Sample | Time Sample | Accession | | | | Normal | Normal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit | Collected | Collected | Number | Test | Result | Units | Range Low | Range High | Flag | |
| | | | | | | | | | | | | _ |
| xx-xxx | XXX | xxxxxxxxx | YYYYMMDD | hh:mm | xxxxxx | xxxxxx | Xxxx | xxxx | xxxx | xxxx | xxxx | |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.8.2
Blood Chemistry - Laboratory Collections
(Safety Population)

Treatment:

| Subject | | | Date Sample | Time Sample | Accession | | | | Normal | Normal | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit | Collected | Collected | Number | Test | Result | Units | Range Low | Range High | Flag |
| xx-xxx | XXX | xxxxxxxxx | YYYYMMDD | hh:mm | xxxxx | xxxxxx | Xxxx | XXXX | xxxx | xxxx | xxxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.8.3
Urinalysis - Laboratory Collections
(Safety Population)

Treatment:

| Subject<br>No. | Sequence | Visit | Date Sample<br>Collected | Time Sample<br>Collected | Accession<br>Number | Test | Result | Units | Normal<br>Range Low | Normal<br>Range High | Flag |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxx | XXX | xxxxxxxxx | YYYYMMDD | hh:mm | xxxxxx | xxxxxx | Xxxx | xxxx | xxxx | xxxx | xxxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine

SAS Program Name: Date:


Neurana 115
Page X of Y

Neurana 115

Listing 16.2.8.4

Drug Screen, Alcohol Screen, Pregnancy, Test Results
(Safety Population)

Treatment:

Subject

| No. | Sequence | Visit Date | Visit | Test | Results |
|--------|----------|------------|----------|---------|-------------|
| xx-xxx | XXX | YYYYMMDD | xxxxxxxx | xxxxxxx | xxxxxxxxxxx |


Neurana 115

Listing 16.2.8.5
Laboratory Values Outside of Normal Range (Safety Population)

Treatment:

| Subject | | | Date Sample | Time Sample | | | | | Normal | Normal | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit | Collected | Collected | Category | Test | Result | Units | Range Low | Range High | Flag |
| xx-xxx | XXX | xxxxxxxxx | YYYYMMDD | hh:mm | xxxxxx | xxxxxx | Xxxx | XXXX | xxxx | xxxx | xxxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name:


Neurana 115

Listing 16.2.8.6.1 Prior Medications (Safety Population)

| Subject No. | Sequence | Visit<br>Date | Medication/<br>Preferred Term/<br>ATC Class | Indication | Dose | Units | Freq | Route | Date Started | Date Stopped |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxx | XXX | YYYYMMDD | xxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxx | xxxxx | xxxx | xxxx | xxxxxx | xxxxxx | YYYYMMDD | YYYYMMDD |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.8.6.2 Concomitant Medications (Safety Population)

Medication/

| Subject | : | Preferred<br>Term/ | | | | | | | | Med Taken |
|---|---|---|---|---|---|---|---|---|---|---|
| No. | Sequence | ATC Class | Indication | Dose | Units Frequency | Route | Date Started | Date Stopped | Ongoing | Due to AE? |
| xx-xxx | XXX | xxxxxxxx/<br>xxxxxxxx/ | xxx | | xxxx | xxxxxx | YYYYMMDD | YYYYMMDD | xxx | xxx |
| | | XXXXXXX | | XXXX | XXXX | | | | | |


Neurana 115

Listing 16.2.8.7.1 Physical Examination (Safety Population)

| Subject | | | | | Other | Physical examination | Abnormal |
|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit Date | Visit | Site | specification | result | Finding |
| xx-xxx | XXX | YYYYMMDD | xxxxxxx | xxxxxxxxx | xxxxxx | Normal/abnormal/not done | xxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

ing 16.2.8.7.2

Listing 16.2.8.7.2 Shift in Physical Examination (Safety Population)

| Subject | | | | | Other | Physical examination | Abnormal |
|---|---|---|---|---|---|---|---|
| No. | Sequence | Visit Date | Visit | Site | specification | result | Finding |
| xx-xxx | XXX | YYYYMMDD | xxxxxxxx | xxxxxxxxxx | xxxxxx | Normal/abnormal/not done | xxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.8.8.1 12-Lead Electrocardiogram Results (Safety Population)

Treatment:

| | | | | | | Ventricular | PR | QRS | QΤ | QTcF |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date of | Time of | Not | | Heart Rate | Interval | Interval | Interval | Interval |
| No. | Sequence | e Assessment | Assessment | Done | Visit | (beats/min) | (msec) | (msec) | (msec) | (msec) |
| · | | | | | | | | | | |
| xx-xxx | XXX | YYYYMMDD | hh:mm | xx | xxxxxx | xxx | xxx | xxx | xxx | xxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine SAS Program Name: Date:


Neurana 115

Listing 16.2.8.8.2 12-Lead Electrocardiogram Assessment (Safety Population)

Treatment:

| Subject<br>No. | Sequence | Visit | Date of ECG | Time of<br>ECG | Clinical<br>Evaluation | Abnormality | Clinical Significance* |
|---|---|---|---|---|---|---|---|
| | | | | | Normal/<br>Abnormal<br>NCS/ | | |
| xx-xxx | XXX | xxxxxxxxx | YYYYMMDD | hh:mm | Abnormal CS | xxxxxxxxx | NCS/CS |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine
\*NCS=not clinically significant, CS=clinically significant.
SAS Program Name:

NOTE TO PROGRAMMER: placebo, 450 mg tolperisone, 30 mg cyclobenzaprine


Neurana 115

Listing 16.2.8.9
Vital Signs
(Safety Population)

Treatment:

| Subject<br>No. | Sequence | Date of Assessment. | Time of<br>Assessment | Not<br>Done | Visit | Time<br>Point | Position | Height (cm) | Weight<br>(kg) | BMI<br>(kg/m^2) | Temperature (C) | Heart<br>Rate (bpm) | Blood<br>Pressure<br>(mm Hg) | Respiration<br>Rate<br>(breaths/min) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxx | XXX | YYYYMMDD | hh:mm | xx | xxxxxx | xxxx | xxxxxx | xx | xx | xx.x | xx | xxx | xxx/xxx | XX |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine

SAS Program Name: Date:


Neurana 115

Listing 16.2.8.10 General Comments (Safety Population)

| Subject | No. Se | equence C | DE | SDTM Domain | Comments |
|---------|--------|-----------|----|-------------|----------|
| xx-x | XX | XXX | xx | xx | xxx |

A=placebo, B=450 mg tolperisone, C=30 mg cyclobenzaprine

SAS Program Name:

Date: